CLINICAL TRIAL: NCT02365571
Title: Single-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Cytochrome P450 Interaction Study of LY3154207 in Healthy Subjects
Brief Title: A Study of LY3154207 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15510; I7S-EW-HBEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-02-17; First posted 2015-02-19 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — LY3154207; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY3154207 (Part A) (Experimental): LY3154207 administered in ascending doses once orally in two of three study periods
  Interventions: Drug: LY3154207
- Placebo (Part A) (Placebo Comparator): Placebo matching LY3154207 administered once orally in one of three study periods.
  Interventions: Drug: Placebo
- LY3154207 (Part B) (Experimental): LY3154207 administered once orally.
  Interventions: Drug: LY3154207
- Placebo (Part B) (Placebo Comparator): Placebo matching LY3154207 administered once orally.
  Interventions: Drug: Placebo
- LY3154207 (Part C) (Experimental): LY3154207 administered once orally on Day 1
  Interventions: Drug: LY3154207
- LY3154207 + Itraconazole (Part C) (Experimental): Itraconazole administered orally (twice daily on Day 3 and then once daily to Day 12). LY3154207 co-administered once orally, on Day 9. Timing and duration of itraconazole dosing may be adjusted based on data from Part A.
  Interventions: Drug: LY3154207; Drug: Itraconazole

INTERVENTIONS:
Drug: LY3154207 — Administered orally
  Arms: LY3154207 (Part A); LY3154207 (Part B); LY3154207 (Part C); LY3154207 + Itraconazole (Part C)
Drug: Placebo — Administered orally
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Itraconazole — Administered orally (twice daily on Day 3 and then once daily to Day 12) as a 10 mg/mL solution
  Arms: LY3154207 + Itraconazole (Part C)

SUMMARY:
This study involves single doses of LY3154207 and will evaluate the effects of LY3154207 on the body. There will be 3 parts to this study.

Part A will test single increasing doses of LY3154207 and will last approximately 7 weeks for each participant. Each participant will receive two doses of LY3154207, if part A is completed.

Part B will test a single dose of LY3154207 and will last approximately 5 weeks for each participant. Part B includes collecting fluid from the spinal column to measure levels of LY3154207.

Part C will include a single dose of LY3154207 given alone and then a second dose given along with itraconazole to look for change in LY3154207 levels. Part C will last about 3 weeks for each participant.

Participants may only enroll in 1 of the 3 parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination
* Female participants not of child-bearing potential
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent
* Have a body mass index (BMI) of 18 to 35 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Part B only: Have medical or surgical conditions in which lumbar puncture is contraindicated
* Part C only: Have known allergy or contraindications to itraconazole

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Up to 48 hours after administration of study drug

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Plasma Part A : Maximum Drug Concentration (Cmax) of LY3154207 | Predose through 48 hours after administration of study drug
Pharmacokinetics (PK) Plasma Part A: Area Under the Concentration Curve (AUC) of LY3154207 | Predose through 48 hours after administration of study drug
Pharmacokinetics (PK) Cerebrospinal Fluid (CSF) Part B: Area Under the Concentration Time Curve (AUC) of LY3154207 | Predose through 48 hours after administration of study drug
Pharmacokinetics (PK) Cerebrospinal Fluid (CSF) Part B: Maximum Drug Concentration (Cmax) of LY3154207 | Predose through 48 hours after administration of study drug
Pharmacokinetics (PK) Plasma Part C: Area Under the Concentration Time Curve (AUC) of LY3154207 when Co-administered with Itraconazole | Predose through 96 hours after administration of study drug
Pharmacokinetics (PK) Plasma Part C: Maximum Drug Concentration (Cmax) of LY3154207 when Co-administered with Itraconazole | Predose through 96 hours after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States